CLINICAL TRIAL: NCT00818363
Title: A Double-Blind, Multi-Center, Placebo-Controlled Trial of SABER-Bupivacaine for Post-Operative Pain Control and Opioid Sparing/Opioid-Related Adverse Event Reduction Following Arthroscopic Shoulder Surgery
Brief Title: A Safety and Effectiveness Study of SABER®-Bupivacaine for Pain Following Shoulder Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C803-017
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; shoulder surgery; opioid
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: SABER-Bupivacaine (Experimental): 5.0 mL SABER-Bupivacaine/Once
  Interventions: Drug: SABER-Bupivacaine
- Group 2: SABER-Placebo (Placebo Comparator): 5.0 mL SABER-Placebo/Once
  Interventions: Drug: SABER-Placebo

INTERVENTIONS:
Drug: SABER-Bupivacaine — Injectable Extended Release Solution; 5.0 mL SABER-Bupivacaine/Once
  Other Names: POSIMIR® bupivacaine solution
  Arms: Group 1: SABER-Bupivacaine
Drug: SABER-Placebo — Injectable Solution; 5.0 mL SABER-Placebo/Once
  Arms: Group 2: SABER-Placebo

SUMMARY:
This is a research study testing SABER-Bupivacaine (an experimental pain-relieving medication). SABER-Bupivacaine is designed to continuously deliver bupivacaine, a common local anesthetic, for a few days in order to treat local post-surgical pain.

The purpose of this study is to investigate safety (if there are any side effects) associated with the use of SABER-Bupivacaine and how well it works in reducing pain and opioid-related side effects following shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to read and understand the consent form, provide written consent, complete trial-related procedures, and communicate with the trial staff.
* Males and females, 18 to 65 years of age, scheduled for shoulder surgery.
* Patients must be healthy or have only mild systemic disease.
* Patients must have ECG wave form within normal limits
* Patients must have blood pressure within normal range.
* Male and female patients must agree to use medically acceptable method of contraception throughout the entire trial period and for 1 week after the trial is completed.
* Patients must refrain from strenuous activities and avoid changes to prescribed exercise levels throughout the course of the trial.

Exclusion Criteria:

* Patients with previous arthroscopic surgery or open surgery on the study shoulder.
* Patients with chronic pain conditions requiring continuous use of corticosteroids for greater than 3 months.
* Patients with fibromyalgia, rheumatoid arthritis, and/or sero-negative inflammatory arthropathies.
* Patients with a below normal calculated creatinine clearance.
* Patients who are pregnant or lactating.
* Patients currently receiving more than 20 mg of hydrocodone daily (or equivalent narcotic dose) on routine basis.
* Patients, who in the Investigator's opinion, have developed opioid tolerance.
* Patients with current or regular use of anticonvulsants, antiepileptics, antidepressants, or monoamine oxidase inhibitors at screening.
* Patients with current or regular use of drugs known to significantly prolong the corrected QT interval
* Patients with known hypersensitivity to local anesthetic agents of the amide type (e.g., lidocaine, bupivacaine).
* Patients with known hypersensitivity to opioids.
* Patients with conditions contraindicated for use of opioids.
* Patients with known or suspected abuse of opioids or other illicit drugs.
* Patients with known or suspected alcohol abuse.
* Participation in another clinical trial at the same time or within 30 days of this trial.
* Patients who, in the Investigator's opinion, should not participate in the trial or may not be capable of following the trial schedule for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Durect
Locations (9):
- Australia (7):
  - Westmead, New South Wales
  - Kippa-Ring, Queensland
  - Adelaide, South Australia
  - Toorak Gardens, South Australia
  - Geelong, Victoria
  - Hampton, Victoria
  - Ringwood East, Victoria
- New Zealand (2):
  - Christchurch
  - Hamilton

REFERENCES:
- [Derived] Hadj A, Hadj A, Hadj A, Rosenfeldt F, Nicholson D, Moodie J, Turner R, Watts R, Fletcher I, Abrouk N, Lissin D. Safety and efficacy of extended-release bupivacaine local anaesthetic in open hernia repair: a randomized controlled trial. ANZ J Surg. 2012 Apr;82(4):251-7. doi: 10.1111/j.1445-2197.2011.05754.x. Epub 2011 Jun 24. PMID 22510183

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Started | 40 | 20
Completed | 40 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (8.8) | 47.6 (9.9) | 47.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 17 | 10 | 27
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.57 (4.17) | 29.33 (5.08) | 27.49 (4.64)

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Intensity on Movement AUC (Time Normalized Area Under the Curve) During the Period 0 to 72 Hours Post-dose.
Description: Mean pain intensity on movement AUC (time normalized area under the curve) during the period 0 to 72 hours post-dose. Subjects assessed their pain intensity using an 11-point Pain Intensity Numeric Rating Scale (PI-NRS) with NRS scores ranging from 0 (no pain) to 10 (worst pain possible). The pain intensity AUC on movement was computed for each subject using the standard trapezoidal rule. For the purpose of better clinical interpretability of the pain AUC, a normalized AUC was computed by dividing it using the time-interval length over which it was computed.
Time Frame: 0 to 72 hours post-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 40 | 20
score on a scale | 5.35 (1.91) | 5.81 (2.25)
Statistical Analysis 1: Comparison: Group 1: SABER-Bupivacaine vs Group 2: SABER-Placebo; Test type: Superiority; p = 0.303, ANCOVA; Includes treatment group and trial site as factors and age as a covariate; LS Mean Difference = -0.64, 95% CI 2-sided [-1.74 to 0.47]

2. Primary Outcome: Supplemental Opioid Use
Description: Mean total morphine-equivalent dose during the period 0 to 72 hours post-dose
Time Frame: 0 to 72 hours post-dose
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 40 | 20
mg | 44.54 (29.62) | 49.94 (45.69)
Statistical Analysis 1: Comparison: Group 1: SABER-Bupivacaine vs Group 2: SABER-Placebo; Test type: Superiority; p = 0.303, ANCOVA; Includes treatment group and trial site as factors and age as a covariate; LS Mean Difference = -10.25, 95% CI 2-sided [-30.04 to 9.55]

3. Secondary Outcome: Number (Frequency) of Participants Reporting Opioid-related Adverse Events
Description: Frequency of subject-reported opioid-related AEs during 0 to 72 hours (0 to 3 days) post-dose and during the trial: constipation, drowsiness, dizziness, nausea, vomiting, respiratory depression, and urinary retention.
Time Frame: 0 to 72 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 40 | 20
Participants
  Day 0 : Constipation | 0 | 0
  Day 0 : Dizziness | 14 | 6
  Day 0 : Drowsiness | 20 | 12
  Day 0 : Nausea | 17 | 11
  Day 0 : Respiratory Depression | 3 | 0
  Day 0 : Urinary Retention | 6 | 1
  Day 0 : Vomiting | 12 | 4
  Day 1 : Constipation | 5 | 1
  Day 1 : Dizziness | 7 | 4
  Day 1 : Drowsiness | 18 | 7
  Day 1 : Nausea | 10 | 5
  Day 1 : Respiratory Depression | 0 | 0
  Day 1 : Urinary Retention | 3 | 2
  Day 1 : Vomiting | 3 | 2
  Day 2 : Constipation | 10 | 5
  Day 2 : Dizziness | 4 | 3
  Day 2 : Drowsiness | 13 | 8
  Day 2 : Nausea | 8 | 2
  Day 2 : Respiratory Depression | 0 | 0
  Day 2 : Urinary Retention | 1 | 1
  Day 2 : Vomiting | 1 | 0
  Day 3 : Constipation | 9 | 4
  Day 3 : Dizziness | 1 | 0
  Day 3 : Drowsiness | 10 | 2
  Day 3 : Nausea | 4 | 1
  Day 3 : Respiratory Depression | 0 | 0
  Day 3 : Urinary Retention | 1 | 0
  Day 3 : Vomiting | 0 | 0

4. Secondary Outcome: Mean Pain Intensity on Movement AUC (Time-normalized AUC) During the Period 0 to 48 Hours Post-dose (0 to 2 Days Post-dose).
Description: Mean pain intensity on movement AUC (time-normalized AUC) during the period 0 to 48 hours post-dose (0 to 2 days post-dose). Subjects assessed their pain intensity using an 11-point Pain Intensity Numeric Rating Scale (PI-NRS) with NRS scores ranging from 0 (no pain) to 10 (worst pain possible). The pain intensity AUC on movement was computed for each subject using the standard trapezoidal rule. For the purpose of better clinical interpretability of the pain AUC, a normalized AUC was computed by dividing it using the time-interval length over which it was computed.
Time Frame: 0 to 48 hours post-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 40 | 20
score on a scale | 5.65 (2.07) | 6.14 (2.23)

5. Secondary Outcome: Supplemental Opioid Use
Description: Mean total morphine-equivalent dose during the period 0 to 48 hours post-dose (0 to 2 days post-dose)
Time Frame: 0 to 48 hours post-dose
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 40 | 20
mg | 37.13 (23.40) | 43.70 (37.44)

6. Secondary Outcome: Time-to-first Use of Opioid Supplemental Pain Medication
Time Frame: 0 to 14 days post-dose
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 40 | 20
hours | 0.43 [0.37 to 0.58] | 0.48 [0.28 to 0.68]

7. Secondary Outcome: Severity of Opioid-related Side Effects
Time Frame: 0 to 14 days post-dose
Population: Severity of opioid related side effects were not collected in the opioid related side effects diary.
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1: SABER-Bupivacaine | Group 2: SABER-Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/20
Other Adverse Events (participants affected / at risk) | 38/40 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SABER-Bupivacaine (N=40) | Group 2: SABER-Placebo (N=20)
Pyrexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SABER-Bupivacaine (N=40) | Group 2: SABER-Placebo (N=20)
Tinnitus (Ear and labyrinth disorders) | 6 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 18 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 4 | 2
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 26 | 15
Vomiting (Gastrointestinal disorders) | 14 | 4
Oedema Peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 1
Sensation Of Pressure (General disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Swelling (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Blood Pressure Increased (Investigations) | 1 | 1
Respiratory Rate Decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 14 | 7
Dysgeusia (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 5 | 4
Hypoaesthesia (Nervous system disorders) | 7 | 3
Paraesthesia (Nervous system disorders) | 9 | 2
Somnolence (Nervous system disorders) | 29 | 16
Dysuria (Renal and urinary disorders) | 8 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes